CLINICAL TRIAL: NCT05020873
Title: Prospective, Observational Study in Sickle Cell Disease Patients on Crizanlizumab Treatment in Middle East Countries and India (SPOTLIGHT)
Brief Title: Prospective, Observational Study in Sickle Cell Disease Patients on Crizanlizumab Treatment in Middle East Countries and India
Acronym: SPOTLIGHT
Status: Terminated | Type: Observational
Why Stopped: sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CSEG101AIC05
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease
Keywords: NIS; sickle cell disease; SCD; crizanlizumab
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — crizanlizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Crizanlizumab: Patients initiated on treatment with commercially available crizanlizumab
  Interventions: Other: Crizanlizumab

INTERVENTIONS:
Other: Crizanlizumab — Prospective observational study. There is no treatment allocation. Patients administered crizanlizumab, that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This is a multicenter, prospective, single-arm observational non-interventional study (NIS), which will be conducted in various countries in the Middle East and India.

DETAILED DESCRIPTION:
The study is designed to collect information on the utilization and effectiveness of crizanlizumab treatment in SCD patients under routine clinical practice conditions, to which the physician has made an independent decision to prescribe crizanlizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with clinical diagnosis of SCD (based on laboratory parameters) of any genotype.
2. Patients newly initiated on treatment with locally approved crizanlizumab.
3. Patients aged 16 years or older at crizanlizumab initiation.

Exclusion Criteria:

1. Patients who did not provide informed consent.
2. Patients who received a stem cell transplant at time of enrollment.
3. Patients who participated in or are participating in a clinical trial at time of enrollment or in the 12 months prior to starting commercial crizanlizumab.
4. According to the investigator's opinion, the patient is an unlikely candidate to provide an accurate medical history and/or to obtain long-term follow-up information for any reasons such as unavailability or severe concomitant illnesses.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with SCD initiated on treatment with commercially available crizanlizumab at sites
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Annualized rate of healthcare visit and home-managed (VOCs) requiring a medical facility visit | 12 months
  The annualized rate of VOCs is defined as the total number of pain crises for a patient occurring from the date of initial infusion with crizanlizumab (commercially available) to the last contact date of the study end date × 365 divided by the number of days during that same time period.
  This calculation accounts for early dropouts or lost to follow-up by extrapolating the VOC rate of every patient to 1 year.

SECONDARY OUTCOMES:
Type of opioids for pain management of healthcare visit and home-managed (VOCs) within the medical facility and at home. | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Type of opioids for pain management of healthcare visit and home-managed (VOCs) within the medical facility and at home to be collected
Dose of opioids for pain management of healthcare visit and home-managed (VOCs) within the medical facility and at home. | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Dose of opioids for pain management of healthcare visit and home-managed (VOCs) within the medical facility and at home to be collected
Duration of use of opioids for pain management of healthcare visit and home-managed (VOCs) within the medical facility and at home. | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Duration of use of opioids for pain management of healthcare visit and home-managed (VOCs) within the medical facility and at home to be collected
Number of healthcare visit and home-managed (VOCs) leading to hospitalization | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Number of healthcare visit and home-managed (VOCs) leading to hospitalization to be collected
Type of healthcare visit and home-managed (VOCs) leading to hospitalization | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Type of healthcare visit and home-managed (VOCs) leading to hospitalization to be collected
Duration of healthcare visit and home-managed (VOCs) leading to hospitalization | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Duration of healthcare visit and home-managed (VOCs) leading to hospitalization to be collected
Outcome of healthcare visit and home-managed (VOCs) leading to hospitalization | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Outcome of healthcare visit and home-managed (VOCs) leading to hospitalization to be collected.
Number of home managed healthcare visit and home-managed (VOCs) as captured in the medical records and as per data from the SCPD-S. | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Number of home managed healthcare visit and home-managed (VOCs) as captured in the medical records and as per data from the SCPD-S to be collected.
  SCPD-S: Sickle Cell Pain Diary - Self Report
Annualized rate home managed healthcare visit and home-managed (VOCs) as captured in the medical records and as per data from the SCPD-S. | month 12 and month 24
  Annualized rate home managed healthcare visit and home-managed (VOCs) as captured in the medical records and as per data from the SCPD-S to be collected.
  SCPD-S: Sickle Cell Pain Diary - Self Report
Percentage of patients free from healthcare visit and home-managed (VOCs) leading to a healthcare visit | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Percentage of patients free from healthcare visit and home-managed (VOCs) leading to a healthcare visit to be collected
Percentage of patients with acute and chronic complications/ end organ damage related to SCD | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Percentage of patients with acute and chronic complications/ end organ damage related to SCD to be collected
Frequency of patients on blood transfusions | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Frequency of patients on blood transfusions to be collected. Blood transfusions: simple/ exchange/ chronic/ episodic
Frequency of patients with SCD-related Healthcare Resource Utilization (HRU) | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Frequency of patients with SCD-related Healthcare Resource Utilization (HRU) to be collected
Number of patients with clinical laboratory parameters abnormalities | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  Number of patients with clinical laboratory parameters abnormalities to be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Novartis Investigative Site, Manama, Bahrain
- Novartis Investigative Site, Al Ahmadi, Kuwait
- Novartis Investigative Site, Doha, Qatar
- Saudi Arabia (2):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jizan

IPD SHARING:
Plan to Share IPD: No